CLINICAL TRIAL: NCT05169164
Title: Observational Cohort Study of Patient Outcomes Following Surgery in Latin American Countries
Brief Title: Latin American Surgical Outcomes Study
Acronym: LASOS
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar MD, PhD, Associate Professor, University of Sao Paulo
Other Study IDs: LASOS
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Complications; Mortality
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: All adult patients (aged 18 years or older) undergoing elective or emergency surgery with a planned overnight stay. No interventions, only observational.
  Interventions: Other: No intervention, observational

INTERVENTIONS:
Other: No intervention, observational — No intervention, observational

SUMMARY:
Methods: International, seven-day observational cohort study of complications following elective or emergency surgery. Objectives: To provide detailed data describing post-operative complications and associated mortality. Number of participants: Our aim is to recruit as many patients from as many hospitals as possible in Latin American nations. Eligible countries for participation: Countries and dependencies in Latin America that are situated in the area stretching from the northern border of Mexico to the southern tip of South America, including the Caribbean. Inclusion criteria: all adult patients aged 18 years or older undergoing elective or emergency surgery during the seven-day study period with a planned overnight stay. Exclusion criteria: patients who are undergoing planned day-case surgery or radiological procedures. Statistical methodology and analysis: Single and multi-level logistic regression models will be constructed to identify factors independently associated with these outcomes and to adjust for differences in confounding factors. A single final analysis is planned at the end of the study. A pre-defined analysis will focus on outcomes of patients who have undergone caesarean section. Study duration: Each nation will select a 7-day period between 1st April and 31th October 2022.

DETAILED DESCRIPTION:
Introduction

More than 310 million patients undergo surgery worldwide each year with reported hospital mortality between 1 and 4%. Recent estimates suggest that 4.2 million deaths occur within 30 days of surgery, and half of these occur in low and middle-income countries (LMIC). Complications are more common and are a leading cause of long-term morbidity and mortality. The International Surgical Outcomes Study (ISOS) confirmed the association between complications and death after surgery at a global scale, but predominantly included high-income nations. More recently, the African Surgical Outcomes Study (ASOS) found that patients undergoing surgery in African nations were twice as likely to die than those in high-income countries (HIC), despite being younger with fewer co-morbid diseases. While there is a global drive to improve access to surgery in LMICs there is a need to implement this safely. Latin America describes a geographic area including 25 nations, and countries within the region have some of the highest income disparity worldwide. Rapid demographic and societal changes have led to an increasing burden of non-communicable disease. Provision of healthcare varies widely within Latin America, with a mix of private, social and government funded schemes. The investigators aim is to conduct a seven-day cohort study of adults undergoing in-patient surgery in Latin America to provide detailed data describing post-operative complications and associated mortality.

Study objectives

Primary objective To evaluate the incidence of 30-day in-hospital complications following elective or emergency in-patient surgery

Secondary objective

* To describe the 30-day in-hospital mortality associated with these complications
* To describe the length of hospital stay
* To describe the pattern of postoperative critical care use
* To describe the effect of postoperative complications on duration of hospital stay
* To describe needs of critical care at postoperative

Primary outcome measure In-hospital post-operative complications of any cause, censored at 30 days following surgery for patients who remain in hospital

Secondary outcome measures

* In-hospital all-cause mortality censored at 30 days following surgery for patients who remain in hospital
* Duration of hospital stay after surgery, censored at 30 days following surgery for patients who remain in hospital
* Admission to critical care within 30 days of surgery during the index admission

Study design

LASOS is an international, observational seven-day cohort study. Data will be collected over a four-month period, each national lead will select seven days over which participating sites within their nation will collect data. The study will take place in Latin American countries and dependencies defined as an area that stretches from the northern border of Mexico to the southern tip of South America, including the Caribbean. All countries and dependencies listed on the page 'Latin America' on Wikipedia as of 16th of September 2019 are eligible to take part. All data collected will be that which is used for routine clinical care in hospital. There will be no additional patient contact.

Study population

Each national group will select a single seven-day period for patient recruitment between 1st April and 31st October 2022. Patients will be identified by the participating sites by review of elective theatre lists, theatre logbooks, handover sheets, emergency admissions and ward lists. All patients undergoing surgery over this period at a hospital taking part in the study will be eligible for inclusion provided the participants meet the following criteria.

Inclusion criteria All adult patients (aged 18 years or older) undergoing elective or emergency surgery with a planned overnight stay.

Surgery is defined as a procedure where a deliberate access to the body is gained via an incision or percutaneous puncture, and where instrumentation is used in addition to the puncture needle, or instrumentation via a natural orifice.

Exclusion criteria Patients who are undergoing planned day-case surgery or radiological procedures.

Risks and benefits

Risks There are no safety considerations relating to the LASOS study. There is no risk of harm to either patients or investigators. The risk of an information governance breach is negligible because no patient identifiable data wil be collected outside each participating hospital.

Benefits

1. to be the driver for improved perioperative care at a policy level in Latin American countries
2. to provide a clear evidence base for further research in the region
3. to provide insights into surgical outcomes that may be applicable to other LMIC settings

Study procedures

Consent procedures Very similar studies have been successfully performed in more than 80 countries. The majority of nations participating in these in prior studies waived the need for informed patient consent, given the dataset includes only those documented as part of routine clinical care and that the data is collected in a fully anonymized format.

Given this precedence, the investigators anticipate that informed consent and ethical approval will not be required for LASOS. The need for consent at each centre will be determined by local coordinators, and a site agreement will be requested from each site lead confirming that data is collected in accordance with local requirements.

Study data

Data will be collected on all eligible patients who undergo surgery during the study week for that country. Centre specific data will be collected at the start of the study period. Standard definitions for all outcomes will be provided to all centres. All relevant study documents will be translated into Spanish, French and Portuguese, and data entry will be available in those languages.

Data collection

Centre specific data will be collected once for each hospital including: university or non-university hospital, number of hospital beds, number of operating rooms, number and level of critical care beds, details about the reimbursement status of the hospital, university hospital status, existence of residency programmes in anaesthesia, surgery, medicine or critical care, availability of a rapid response team, if the hospital holds valid accreditation (ONA, Qumentum or Joint Commission) and the ratio of nursing staff to hospital beds in post-operative care areas.

Data will be collected in individual hospitals on a paper CRF for each patient recruited. Paper CRFs will be stored within a locked office in each centre. This will include identifiable patient data in order to allow follow-up of clinical outcomes. The CRF will be completed for all participants, with separate data collection for patients having a caesarean section.

Data will be anonymized by generating a unique numeric code ('LASOS ID') and transcribed by local investigators onto an internet based electronic CRF. Patients will only be identified on the electronic CRF by their LASOS ID. A patient list will be used in each centre to match the LASOS ID to individual patients in order to record clinical outcomes and supply any missing data points. Once the local coordinator confirms data entry is complete for their hospital the coordinators will receive a spreadsheet of raw (un-cleaned) data, allowing further checks for data completeness and accuracy.

Study group organization

LASOS will be led by the study management group who will be responsible for study administration, communication between project partners, data collation and data management. National coordinators will lead the project in each nation and:

* Identify local coordinators in participating hospitals
* Assist with translation of study paperwork as required
* Ensure distribution of study paperwork and other materials
* Ensure necessary regulatory approvals are in place prior to the start date
* Ensure good communication with the participating sites in his/her nation

Local coordinators in individual institutions will have the following responsibilities:

* Provide leadership for the study in their institution
* Ensure all relevant regulatory approvals are in place for their institution
* Ensure adequate training of all relevant staff prior to data collection
* Supervise daily data collection and assist with problem solving
* Act as guarantor for the integrity and quality of data collected
* Ensure timely completion of eCRFs by supervising local data entry
* Communicate with the relevant national coordinator
* Review and sign data sharing agreement at time of site opening.

End of study definition

The end of the study is defined as the end of the 30-day follow-up for the last patient included. Data analysis will follow this.

Statistical considerations

Sample size All eligible patients during the recruitment period will be included. The investigators do not have a specific sample size and statistical models will be adapted to the event rate provided by the sample recruited.

Statistical analysis No comparison will be made between individual nations and all national and institutional level data will be anonymized prior to publication. Categorical variables will be described as proportions. Continuous variables will be described as mean and standard deviation, if normally distributed, or median and inter-quartile range, if not normally distributed.

Univariate analysis will be performed to test factors associated with post-operative complications, admission to critical care and in-hospital death. Single-level and hierarchical multi-level logistic regression models will be constructed to identify factors independently associated with these outcomes and to adjust for differences in confounding factors. Factors will be entered into the models based on biological plausibility and low rate of missing data. Results of logistic regression will be reported as adjusted odds ratios (OR) with 95% confidence intervals. The models will be assessed in sensitivity analyses to explore possible interacting factors and examine any effect on the results. Imputation will be considered for important missing variables. A single final analysis is planned at the end of the study.

A pre-specified, separate analysis will be performed restricted to patients undergoing caesarean section as this group have previously been identified as having very poor outcomes compared to mothers in HIC.

Ethics

It is anticipated that requirements at participating nations will vary. This will vary by nation and the study will be conducted in line with local legal and regulatory requirements. In prior studies of this design across more than 80 countries, the vast majority of nations have been happy to proceed without individual patient level consent. It is the national and local investigators responsibility to clarify the need for ethics or other regulatory approvals, and for ensuring these are in place prior to data collection. Centres will not be permitted to record data without providing confirmation that the necessary ethics or other regulatory approvals are in place.

The investigators will ensure that this study is conducted in accordance with the Principles of the Declaration of Helsinki as amended in Tokyo (1975), Venice (1983), Hong Kong (1989), South Africa (1996), Edinburgh (2000), Washington DC (2002), Tokyo (2004), Seoul (2008) and Fortaleza (2013) as described at the following internet site: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects.

Data handling and record keeping

Data management Data will be recorded on paper CRFs and uploaded onto the study database where only anonymized data is collected. Each centre will also maintain an investigator site file including a protocol, local investigator delegation log, CRFs, documentation of the relevant regulatory approvals if applicable, screening log and patient list. The study specific documents will be available to download on the LASOS study website. LASOS CRFs will be stored securely in a locked cupboard and handled only by clinical staff familiar with handling personal data.

Source data Since only routine clinical data is collected, the study CRFs will be completed based on the hospital medical records, which are considered as source data for this study.

Confidentiality All identifiable data collected, processed and stored for the purposes of the project will remain confidential at all times and comply with Data Protection Act, the General Data Protection Regulation (GDPR), NHS Caldecott Principles, the UK Policy Framework for Health and Social Care Research. Data will be collected by the patients' direct care team and will be anonymized prior to transfer to the LASOS study management group. Access to the data entry system will be protected by username and password, delivered during the registration process for individual local investigators. All electronic data transfer between participating centres and the coordinating centre will be encrypted using the SSL 3.0 protocol (HTTPS). Desktop and laptop security will be maintained through usernames and passwords. The datacentre facilities are accredited to robust international standards that are standard for transfer of healthcare data: ISO 27001, ISO 9001, ISO 14001 and PCI DSS. At time of registration on the database entry portal, all users will review an information governance document and electronically sign to confirm that the centre will abide by it. Individual site data sharing agreements will be requested from the local coordinator.

Record retention and archiving All trial documentation and data will be stored for two years after the main study findings are publicly reported, and then archived or destroyed by participating hospitals according to local hospital policies. Electronic data sets will be stored indefinitely.

Data management and ownership In line with the principles of data preservation and sharing, the steering committee will, after publication of the overall dataset, consider all reasonable requests to conduct secondary analyses. The primary consideration for such decisions will be the quality and validity of any proposed analysis. Only summary data will be presented publicly and all national, institutional and patient level data will be strictly anonymized. Individual patient data provided by participating hospitals remain the property of the respective institution. Once each local coordinator has confirmed the data provided from their hospital are both complete and accurate, the centre will be provided with a spreadsheet of the raw (un-cleaned) data for their hospital. The complete LASOS dataset, anonymized with respect to participating patients, hospitals and nations, will be made freely and publicly available two years following publication of the main scientific report. Prior to this, the steering committee is not under any obligation to release data to any collaborator or third party if the steering committee believe this is not in keeping with the wider aims of the LASOS project.

Safety reporting

The trial involves negligible risks to patients and investigators, as it involves only collection of anonymized routinely collected data. Adverse events will not be monitored or reported.

ELIGIBILITY:
Inclusion Criteria:

All adult patients (aged 18 years or older) undergoing elective or emergency surgery with a planned overnight stay.

Surgery is defined as a procedure where a deliberate access to the body is gained via an incision or percutaneous puncture, and where instrumentation is used in addition to the puncture needle, or instrumentation via a natural orifice.

Exclusion Criteria:

Patients who are undergoing planned day-case surgery or radiological procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Each national group will select a single seven-day period for patient recruitment between 1st April and 31st October 2022. Patients will be identified by the participating sites by review of elective theatre lists, theatre logbooks, handover sheets, emergency admissions and ward lists. All patients undergoing surgery over this period at a hospital taking part in the study will be eligible for inclusion provided they meet the following criteria.
Sampling Method: Non-Probability Sample
Enrollment: 23000 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  In-hospital postoperative complications of any cause, censored at 30 days following surgery for patients who remain in hospital

SECONDARY OUTCOMES:
Mortality | 30 days
  In-hospital all-cause mortality censored at 30 days following surgery for patients who remain in hospital
Hospital stay | 30 days
  Duration of hospital stay after surgery, censored at 30 days following surgery for patients who remain in hospital
Critical care | 30 days
  Admission to critical care within 30 days of surgery during the index admission

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila Hajjar, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Banco de Prótesis, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Undecided
In line with the principles of data preservation and sharing, the steering committee will, after publication of the overall dataset, consider all reasonable requests to conduct secondary analyses. Only summary data will be presented publicly and all national, institutional and patient level data will be strictly anonymised. Individual patient data provided by participating hospitals remain the property of the respective institution. The complete LASOS dataset, anonymised with respect to participating patients, hospitals and nations, will be made freely and publicly available two years following publication of the main scientific report.

REFERENCES:
- [Derived] Latin American Surgical Outcomes Study (LASOS) group. Patient outcomes after surgery in 17 Latin American countries (LASOS): a 7 day prospective cohort study. Lancet Glob Health. 2025 Apr;13(4):e635-e645. doi: 10.1016/S2214-109X(24)00558-8. PMID 40155102
- [Derived] Hajjar LA, Quintao VC, Vieira APZ, Nakada LN, Pearse RM, Ramirez MBD, la Medina AR, Alvarez A, McLoghlin S, Boccalatte L, Padmore G, Feraudy I, Martinez M, Villablanca N, Perez C, Calvache JA, Lincango E, Sosa R, Shu S, Riva J, Godinez L, Frias M, Major D, Licea M, Batista S, Charles S, Vaca M, Rosado ID, Borunda D, Zaky OB, Cardona CMC, Carmona MJC, Stefani LC. Latin American surgical outcomes study: study protocol for a multicentre international observational cohort study of patient outcomes after surgery in Latin American countries. BJA Open. 2022 Aug 19;3:100030. doi: 10.1016/j.bjao.2022.100030. eCollection 2022 Sep. PMID 37588582
- See also: Study Principal Web-site — http://lasos-study.org